CLINICAL TRIAL: NCT00048386
Title: A Pilot Study of Gene Modified Autologous Neuroblastoma Vaccine for the Post-Chemotherapy Treatment of High-Risk Neuroblastoma
Brief Title: Neuroblastoma Vaccine for Treatment of High-Risk Neuroblastoma After Chemotherapy
Acronym: CYCHE2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Malcolm Brenner (Other)
Collaborators: Baylor College of Medicine (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Malcolm Brenner, Professor Departments of Medicine and Pediatrics/Director Center for Cell and Gene Therapy, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H8354; HIGH RISK NEUROBLASTOMA
Record Dates: First submitted 2002-10-30; First posted 2002-11-01 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: autologous neuroblastoma vaccine — A vaccine dose of 0.3 x 108 IL-2 secreting cells/patient/injection will be used. Injections will be given twice monthly for two months, then monthly for four months, for a total of eight vaccine injections over six months.

SUMMARY:
PRIMARY OBJECTIVE To determine the percentage of patients with high risk neuroblastoma in first or subsequent partial response or better, or with microscopic residual bone marrow disease, who demonstrate an immunological anti-tumor response at any time during, and for up to 12 months from initiation of, treatment with subcutaneous injections of autologous neuroblastoma cells, genetically modified by adenoviral vectors to secrete interleukin-2 (IL-2) (autologous neuroblastoma vaccine)

SECONDARY OBJECTIVES 1. To determine the toxicity of the autologous neuroblastoma vaccine given according to this schedule 2. To obtain preliminary data on the effect of vaccine administration on progression-free survival from high-risk neuroblastoma

DETAILED DESCRIPTION:
Tumor cells from subjects with high-risk neuroblastoma will be obtained at the time of presentation and initial diagnosis, during routine surveillance of bone marrow disease status, or at the time of surgical resection of disease during primary chemotherapy. The tumor cells will be irradiated to prevent the possibility of tumor growth. Autologous neuroblastoma tumor cells will be used to treat neuroblastoma following the completion of primary or salvage chemotherapy when peripheral blood lymphocyte counts have recovered to > 500 CD3+ cells/mm3. This preceding chemotherapy may or may not have included bone marrow or peripheral stem cell rescue. Therefore, following the achievement of best response with chemotherapy, vaccine will be administered for 6 months. Vaccine modified for secretion of IL-2 will be used.

Vaccine therapy will commence after complete recovery from the side effects of primary or salvage chemotherapy, as long as the subject has an absolute CD3+ lymphocyte count and an absolute neutrophil count greater than 500/mm3. A vaccine consisting of 0.3 x 10 8 cells/patient will be given per injection, based on data from the Phase I studies. Injections will be given twice monthly for two months, then monthly for four months, for a total of eight vaccine injections over six months. The immune effects of the vaccine, toxicity of treatment, and anti-tumor effects will be periodically assessed. Further evaluation will be done annually.

The first and second vaccine injection sites will be "punch biopsied" one week after the injection. Several x-rays and various types of scans will also be taken to assist with monitoring the status of the neuroblastoma. Complete details of the evaluations required by this study are included in.

Subjects may receive supportive care for any acute or chronic toxicity from the injections, including blood product support, antibiotics, and other appropriate intervention. Pneumocystis carinii prophylaxis initiated during chemotherapy may be continued during vaccine therapy for as long as deemed appropriate by the investigator. As well, subjects may receive concurrent therapy with cis-retinoic acid at the discretion of the treating physician.

An adenoviral vector is being used to transduce the cells ex-vivo. Subjects will not be treated with the viral vector.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients with high risk neuroblastoma defined below, who, following completion of front-line or salvage chemotherapy that may or may not have included high-dose chemotherapy followed by peripheral blood stem cell or bone marrow rescue with or without cis-retinoic acid, have achieved partial response or better, or who have microscopic residual bone marrow:

  1. INSS Stage 4 neuroblastoma, diagnosed between 1 and 21 years of age (inclusive)
  2. INSS Stage 3, N-myc amplified neuroblastoma, diagnosed between 1 and 21 years of age (inclusive)
  3. INSS Stage 3, N-myc non-amplified, Shimada unfavorable histology neuroblastoma, diagnosed between 1 and 21 years of age (inclusive)
  4. INSS Stages 2A or 2B, N-myc amplified, Shimada unfavorable histology, diagnosed between 1 and 21 years of age (inclusive)
  5. INSS Stage 4 neuroblastoma, with Shimada unfavorable histology, diagnosed under 365 days of age
* Patients with intermediate or low risk neuroblastoma, who have achieved a second or subsequent partial response or better following chemotherapy treatment of first or subsequent relapse
* Patients must have recovered from the toxic effects of prior chemotherapy prior to treatment on this study, and must have both an absolute lymphocyte count and an absolute neutrophil count greater than 500/mm3.
* Patients with disease status outlined in the first bullet who have been treated with allogeneic tumor vaccine are eligible for treatment with autologous tumor vaccine when that product becomes available
* Patients may not concurrently receive any investigational agents or other tumor vaccines.
* Patients must be HIV-negative.
* Female patients must not be pregnant or lactating.
* Patients must have autologous transduced neuroblastoma cells available that are demonstrably producing > 150 pg IL-2/10e6 cells/24 hours.
* Patients or legal guardians must sign an informed consent according to institutional guidelines.
* Patients who are sexually active must be willing to utilize one of the more effective birth control methods during the study and for 3 months after the study is concluded. The male partner should use a condom.

Max Age: 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 1999-11; Primary Completion 2004-12 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Patients who demonstrate immunological anti-tumor response at any time during, and for up to 12 months from initiation of, treatment with injections of autologous neuroblastoma cells, genetically modified by adenoviral vectors to secrete IL-2 | 12 months post injections

SECONDARY OUTCOMES:
To determine the toxicity of the autologous neuroblastoma vaccine given according to this schedule | 15 years
To obtain preliminary data on progression-free survival from high-risk neuroblastoma following vaccine administration | 15 years

CONTACTS AND LOCATIONS:
Overall Officials: Heidi V Russell, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States